CLINICAL TRIAL: NCT01002430
Title: Endocardial VEGF-D Gene Therapy for the Treatment of Severe Coronary Heart Disease - A Phase 1 Single-blinded Placebo-controlled Phase 1 Clinical Trial
Brief Title: EndocardialVascularEndothelialGrowth Factor D(VEGF-D)Gene Therapy for the Treatment of Severe Coronary Heart Disease
Acronym: KAT301
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Juha Hartikainen, Professor, Director, Heart Center, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5101035
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Angina Pectoris; Myocardial Infarction
Keywords: Myocardial ischemia; Refractory angina pectoris; Vascular endothelial growth factor; Gene therapy; Perfusion
MeSH Terms: conditions — Angina Pectoris; Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gene therapy (Experimental)
  Interventions: Biological: VEGF-D gene transfer
- Control (No Intervention): Control patients will have electroanatomic mapping procedure but no gene injections.

INTERVENTIONS:
Biological: VEGF-D gene transfer — Gene transfer will be performed by using endocardial injection system (NOGATM) and an escalating dose of 1x109, 1x1010 and 1x1011 vpu of AdVEGF-D will be injected into 10 sites of the myocardium (0.2 ml per site).
  Arms: Gene therapy

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of catheter mediated endocardial adenovirus VEGF-D gene therapy in patients with severe coronary heart disease.

DETAILED DESCRIPTION:
Study objective(s):

The purpose of the study is to evaluate the safety and efficacy of catheter mediated endocardial adenovirus VEGF-D gene transfer in patients with severe coronary heart disease to whom revascularisation cannot be performed ("no option -patients"). The primary objective is safety of the gene therapy and the secondary objective is the efficacy of gene therapy to improve myocardial perfusion as measured by MRI, PET and left ventricular function as measured by echocardiography as well as to improve functional status as measured by bicycle ergometer test. Quality of life will be monitored with a personal interview and the consumption of nitrate medication.

Study design:

This is a randomised, single-blinded, placebo controlled single centre Phase I study for patients with coronary heart disease to whom no other treatment than standard medication is available. Patients will be randomized 4:1 to the treatment group and control group. Control patients will not be treated with gene injections but only with cardiac electroanatomical mapping.

Study population:

Up to thirty patients will be recruited from the area of Kuopio University Hospital in the study. The patients will be selected for the trial on the basis of coronary angiogram imaging. Only those patients who are not eligible for the coronary angioplasty or bypass operation ("no option -patients") due to diffuse coronary stenosis, small coronary vessels, repeated revascularisation or too high risk for operation, will be included.

Assessments:

Assessments for safety are recording of adverse events (Appendix 4), laboratory assessments and transthoracic echocardiography. Assessments for efficacy are clinical symptoms and need for nitrate medication, cardiac MRI, PET and bicycle ergometer test. Other assessments are 24-hour Holter recording, transthoracal echocardiography, quality of life and PCR reactions for the detection of gene and virus vector.

Investigational drug product:

First generation replication-deficient AdVEGF-D produced in 293 cells (refer to product master file (PMF-VD-08-001)) will be injected into ten sites in the endocardium. In the beginning, an escalating dose of 1x109, 1x1010 and 1x1011 vpu of virus in a total volume of 2 ml (10 times 0.2 ml) will be used. On the basis of fifteen patients an interim analysis will be performed to evaluate the most suitable dose of virus which will be used for the rest of the study patients. Control patients will not be treated with drug product, only electroanatomical mapping will be performed.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed,
* age between 30 and 80 years,
* significant angina pectoris (CCS II-III) despite of maximal medication,
* significant stenosis in coronary angiography (stenosis > 60 %),
* contraindication to coronary angioplasty or by pass operation (diffuse or distal stenosis,
* chronic total occlusion,
* vessels with difficult anatomy,
* stenosis with severe calcifications,
* stenosis in small vessels (< 2.5 mm)),
* reversible myocardial perfusion defects detected by pharmacological adenosine or dobutamine assisted perfusion MRI,
* angina pectoris or ischemic ST-depression (> 1 mm) in the exercise test,
* left ventricle wall > 8 mm detected by transthoracal echocardiography (treatment area).

Exclusion Criteria:

* women in fertile age,
* patients with type 1 diabetes mellitus or severe end-stage type 2 diabetes mellitus,
* diabetic retinopathy,
* atrial fibrillation,
* clinically significant anemia (hemoglobin count < 120 mg/l in male, < 110 mg/l in female; hematocrit < 0.36), leukopenia (b-leukocyte count < 3.0x109/l), leukocytosis (b-leukocyte count > 12.0x109/l) or thrombocytopenia (b-thrombocyte count < 100x109/l), renal insufficiency (s-creatinine > 160mg/l),
* liver insufficiency (s-alanine amino transferase and s-alcaline phosphatase over 2 x normal),
* haematuria of unknown origin,
* severe hypertension (systolic blood pressure > 200 mmHg or diastolic blood pressure > 110 mmHg) or significant hypotension (systolic blood pressure < 90mmHg),
* significant obesity (BMI > 35),
* cardiac pacemaker,
* acute infection,
* immunosuppressive medication,
* significant impairment of the left ventricular function (EF < 25% in TTE or CO < 2 l in MRI),
* congestive heart failure,
* haemodynamically significant (gradus 3-4/4) aortic regurgitation or other heart disease needing surgery,
* recent ( < 6 weeks) acute coronary syndrome or myocardial infarction (elevated CK-MB or cardiac troponin),
* PCI or CABG or TIA/stroke,
* previous or current malignancy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-01-10 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2015-06-15 (Actual)

PRIMARY OUTCOMES:
Assessments for safety and tolerability as measured as the acute and late adverse effects, laboratory parameters, biodistribution of the vector, anti-adenovirus antibodies and VEGF-levels before and in several time points after the gene transfer. | 1 year

SECONDARY OUTCOMES:
Efficacy of GT to increase myocardial perfusion in MRI and PET. | 1 year
Functional capacity in exercise test, LV-function in echocardiography, arrhythmias in 24-hours Holter-recording will be analyzed. | 1 year
Improvement in symptoms, QOL and medication. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Juha Hartikainen, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Derived] Leikas AJ, Hassinen I, Kivela A, Hedman A, Mussalo H, Yla-Herttuala S, Hartikainen JEK. Intramyocardial adenoviral vascular endothelial growth factor-D∆N∆C gene therapy does not induce ventricular arrhythmias. J Gene Med. 2022 Aug;24(8):e3437. doi: 10.1002/jgm.3437. Epub 2022 Jul 6. PMID 35750637